CLINICAL TRIAL: NCT05067426
Title: The 10/7 HIIT Shock Cycle Study: The Effects of a 7-Day High-Intensity-Interval Training Shock Microcycle on Endurance Performance, Well-Being, Stress and Recovery in Endurance Trained Athletes - Randomized Controlled Trial
Brief Title: The 10/7 HIIT Shock Cycle Study: Effectiveness of 10 HIIT Sessions in 7 Days
Acronym: THESIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salzburg (Other)
Collaborators: Paracelsus Medical University (Other); Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Nils Haller, PhD, Senior Researcher, University of Salzburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHaller
Record Dates: First submitted 2021-09-06; First posted 2021-10-05 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Athlete; Performance
Keywords: High-intensity interval training; Microcycle; Endurance training; Load monitoring; Athlete performance; HIT training; Block training; HIT block; Polarized training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in either one of 2 intervention groups or a control group (ratio 1:1:1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT-HV (Experimental): HIIT-HV - high intensity interval training high volume
  Participants complete a total of 10 HIIT sessions over a 7-day period consisting of 5 x 4-minute intervals at an intensity of 90-95% of their individual maximum heart rate (HRmax), interspersed with a 2.5-minute active recovery period. Each training session is followed by 30 minutes of low-intensity training (total of 300 minutes of additional low-intensity training during this period).
  Interventions: Other: Exercise
- HIIT-LV (Experimental): HIIT- LV - high intensity interval training low volume
  Participants complete a total of 10 HIIT sessions over a 7-day period consisting of 5 x 4-minute intervals at an intensity of 90-95% of their individual maximum heart rate (HRmax), interspersed with a 2.5-minute active recovery period.
  Interventions: Other: Exercise
- Control group (No Intervention): Participants continue with their regular training program.

INTERVENTIONS:
Other: Exercise — high-intensity interval training sessions
  Arms: HIIT-HV; HIIT-LV

SUMMARY:
A randomized, controlled trial to evaluate the effects of two versions of 10 high intensity interval trainings (HIIT) within a 7-day shock microcycle on endurance performance, well-being, health, stress and recovery in trained athletes.

DETAILED DESCRIPTION:
Thirty-six trained endurance athletes will be recruited and randomly assigned to either a "high volume (HIIT-HV)" group, a "low volume (HIIT-LV)" group, or a control group. All participants will be monitored before (9 days), during (7 days), and after (14 days) a 7-day training intervention, for 30 days. Participants in both intervention groups will complete 10 HIIT sessions within the period of 7 days, with an additional 30 minutes of low-intensity training exclusively in HIIT-HV. HIIT sessions consist of aerobic HIIT, i.e., 5x4min at 90-95% of maximal heart rate interspersed by 2.5 min active recovery periods. To determine the effects of the intervention, performance diagnostics, and a 5 kilometer time trial will be conducted before and after the intervention. In addition, participants are closely monitored for general health, stress, fatigue, recovery, neuromuscular performance, executive functions and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* aged 18-45 years
* Proof of physical fitness (e.g. sports medical examination required) for measurements with higher intensities (e.g. endurance tests, competition simulation)
* Competition experience at the national or international level in an endurance sport
* VO2max ≥50ml/kg/min for females; ≥55 ml/kg/min for males or a 5-kilometer (km) time trial performance of ≤ 20:00 min (female), or ≤ 18:30 min (male)

Exclusion Criteria:

* Systemic disease or other known pathology in the organs: heart, lungs, kidney, stomach, spleen, liver, gall bladder, and intestines.
* Evidence of pulmonary disease: forced expiratory volume in one second/forced expiratory volume < 70% with/without symptoms (cough, sputum) or other evidence of pulmonologic disease.
* Diabetes II.
* Neurological or psychological disease of any kind.
* Currently undergoing medical or psycho-therapeutic treatment.
* Health condition that does not allow regular participation in the training forms (e.g. acute illnesses such as fever or other flu-like infections within the last 7 days before the start of the study), orthopedic diseases, injuries to the muscular, bone, joint or tendon apparatus within the last three months.
* Alcohol or drug abuse.
* Already high training volume with high intensity training (more than 2 weekly training sessions of high-intensity training)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Endurance performance I | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of maximal oxygen uptake (VO2max in ml/min/kg) compared to baseline and group
Endurance performance II | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of peak performance (Ppeak in Watt) compared to baseline and group
Endurance performance III | 20 to 22 days (the assessment is conducted once before, and once after the intervention)
  Change of 5 kilometer time trial performance (in sec) compared to baseline and group
Endurance performance IV | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of lactate threshold (in km/h) compared to baseline and group
Endurance performance V | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of ventilatory thresholds (in km/h) compared to baseline and group
Endurance performance VI | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of running economy (in ml/min/kg) compared to baseline and group

SECONDARY OUTCOMES:
Change of questionnaire scores - well-being | 30 days (questionnaires will be given to participants several times before, during, and after the intervention.)
  Change of questionnaire scores compared to baseline and group as determined by a Visual-Analogue-Scale (from 0-100 millimeters). Higher scores indicate poorer well-being.
Change of questionnaire scores - muscular fatigue | 30 days (questionnaires will be given to participants several times before, during, and after the intervention.)
  Change of questionnaire scores compared to baseline and group as determined by a Visual-Analogue-Scale (from 0-100 millimeters). Higher scores indicate higher degree of fatigue.
Change of questionnaire scores - vitality | 30 days (questionnaires will be given to participants several times before, during, and after the intervention.)
  Change of questionnaire scores compared to baseline and group as determined by a Likert-Scale (from 0-10). Higher scores indicate higher vitality.
Change of questionnaire scores - rate of fatigue | 30 days (questionnaires will be given to participants several times before, during, and after the intervention.)
  Change of questionnaire scores compared to baseline and group as determined by a Likert-Scale (from 0-10). Higher scores indicate higher degree of fatigue.
Change of questionnaire scores - sleep quality | 30 days (questionnaires will be given to participants several times before, during, and after the intervention.)
  Change of questionnaire scores compared to baseline and group as determined by a Likert-Scale (from 1-7). Higher scores indicate poorer sleep.
Change of blood count | 30 days (blood is drawn from participants several times before, during, and after the intervention.)
  Change of blood count concentrations compared to baseline and group
Change of cell-free DNA | 30 days (blood is drawn from participants several times before, during, and after the intervention.)
  Change of cell-free DNA concentrations compared to baseline and group
Change of creatine kinase | 30 days (blood is drawn from participants several times before, during, and after the intervention.)
  Change of creatine kinase concentrations compared to baseline and group
Change of urea | 30 days (blood is drawn from participants several times before, during, and after the intervention.)
  Change of urea concentrations compared to baseline and group
Change of blood lactate | 30 days (blood is drawn from participants several times before, during, and after the intervention.)
  Change of blood lactate concentrations compared to baseline and group
Change of cytokines | 30 days (blood is drawn from participants several times before, during, and after the intervention.)
  Change of cytokine concentrations compared to baseline and group
Change of miRNA | 30 days (blood is drawn from participants several times before, during, and after the intervention.)
  Change of miRNA compared to baseline and group
Change of neuromuscular performance | 30 days (neuromuscular performance is assessed several times before, during, and after the intervention)
  Change of neuromuscular performance (counter movement jump height in cm) measured on a contact plate (AMTI, Watertown, USA) compared to baseline and group
Change of body weight | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of body weight in kg compared to baseline and group
Change of fat free mass | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of fat free mass in kg compared to baseline and group
Change of fat mass | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of fat mass in kg compared to baseline and group
Change of forced expiratory volume | 10 to 21 days (assessment is conducted once before the intervention and repeated three times afterwards, i.e. 3, 7 and 14 days after the completion of the intervention)
  Change of forced expiratory volume in liters compared to baseline and group
Change of power output during exercise | 7 days
  Change of power output in Watt (as determined via Stryd, Boulder, USA) during the intervention compared to baseline and group
Change of sleep quality I - GPS watch | 30 days (sleep is assessed several times before, during, and after the intervention)
  Change of sleep quality compared to baseline and group as determined by a GPS (Global Positioning System) watch
Change of sleep quality II - ABIOS App | 30 days (sleep is assessed several times before, during, and after the intervention)
  Change of sleep quality compared to baseline and group as determined by the ABIOS (Algorithmik Biodata System) application
Correlations between sleep quality devices | 30 days
  To determine the correlations between different sleep monitoring devices, i.e. the GPS watch (see outcome 27), the ABIOS system (see outcome 28) and the sleep quality questionnaire (see outcome 11)
Change of parameters recorded by an electrocardiogram - mean heart rate | 30 days (an electrocardiogram is written several times before, during, and after the intervention)
  Change of mean heart rate compared to baseline and group
Change of parameters recorded by an electrocardiogram - heart rate variability | 30 days (an electrocardiogram is written several times before, during, and after the intervention)
  Change of heart rate variability (root mean sum of squared distance in ms) compared to baseline and group
Change of executive functions - Eriksen flanker task | 30 days (executive functions are tested several times before, during, and after the intervention)
  Change of executive functions compared to baseline and group. This is recorded through a modified Eriksen flanker task consisting of 108 images showing five white arrows on a black screen.
Change of executive functions - 2 back task | 30 days (executive functions are tested several times before, during, and after the intervention)
  Change of executive functions compared to baseline and group. This is assessed through a 2-back task showing dots on a dice, numbers and geometrical figures.
Cardiac ultrasound | 1 day (this outcome will be determined once before study start)
  Description of an athlete cohort regarding cardiac chamber volume (in ml, determined via EPIQ CVX, X5-1, Philips Healthcare, Andover, MA, USA)
Adherence to training program | 7 days
  Adherence to the HIIT training programs (determined as the ratio of training sessions performed to prescribed training sessions). This is determined by the researchers by checking the training data of the athletes. For example, if 9 out of 10 sessions were performed, this means 90% adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Stoeggl, Professor, PhD, Study Chair — University of Salzburg
Locations (1):
- University of Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomaskovic A, Strepp T, Stoggl TL, Neuberger EWI, Simon P, Haller N. Acute and Chronic Effects of a High-Intensity Interval Training Shock Microcycle on Cell-Free DNA: A Randomized Controlled Trial. Sports Med Open. 2025 Nov 21;11(1):132. doi: 10.1186/s40798-025-00923-9. PMID 41269434
- [Derived] Strepp T, Blumkaitis JC, Sareban M, Stoggl TL, Haller N. Training Intensity Distribution of a 7-Day HIIT Shock Microcycle: Is Time in the "Red Zone" Crucial for Maximizing Endurance Performance? A Randomized Controlled Trial. Sports Med Open. 2024 Sep 5;10(1):97. doi: 10.1186/s40798-024-00761-1. PMID 39235639
- [Derived] Strepp T, Blumkaitis JC, Haller N, Stoggl TL. Adding LIT to HIIT: Is Low-Intensity Training Vital for Endurance-Trained Athletes during a 7-day HIIT Shock Microcycle? Med Sci Sports Exerc. 2024 Aug 1;56(8):1408-1421. doi: 10.1249/MSS.0000000000003435. Epub 2024 Apr 6. PMID 38587921
- [Derived] Stoggl TL, Blumkaitis JC, Strepp T, Sareban M, Simon P, Neuberger EWI, Finkenzeller T, Nunes N, Aglas L, Haller N. The Salzburg 10/7 HIIT shock cycle study: the effects of a 7-day high-intensity interval training shock microcycle with or without additional low-intensity training on endurance performance, well-being, stress and recovery in endurance trained athletes-study protocol of a randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 May 7;14(1):84. doi: 10.1186/s13102-022-00456-8. PMID 35526065